CLINICAL TRIAL: NCT01230424
Title: Effect of Intra-articular Steroids on Structural Progression of Knee OA: A Randomized Controlled Trial
Brief Title: Effect of Steroid Injections in a Knee With Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIH NIAMS R01-AR057802; Tufts MC IRB Protocol # 9417 (Other: Tufts Medical Center)
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: OA; Knee arthritis; MRI; Steroid
MeSH Terms: conditions — Osteoarthritis | interventions — Triamcinolone Acetonide; Sodium Chloride; Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triamcinolone Acetonide (Experimental): 40 mg into the study knee joint every 12 weeks for a total of 8 injections.
  Interventions: Drug: Triamcinolone Acetonide
- Sodium Chloride (Placebo Comparator): 0.9% Sodium chloride injection as Placebo will be given into the study knee once every 12 weeks for a total of 8 injections.
  Interventions: Drug: 0.9% Sodium Chloride Injection as Placebo

INTERVENTIONS:
Drug: Triamcinolone Acetonide — 40 mg into the study knee joint every 12 weeks for a total of 8 injections.
  Other Names: Kenalog
  Arms: Triamcinolone Acetonide
Drug: 0.9% Sodium Chloride Injection as Placebo — Sodium chloride injection will be given into the study knee once every 12 weeks for a total of 8 injections.
  Other Names: Normal Saline for injection
  Arms: Sodium Chloride

SUMMARY:
A steroid (triamcinolone) 40 mg will be compared to placebo in a randomized placebo-controlled clinical trial testing the effect of this steroid versus placebo given into the study knee joint that has osteoarthritis (OA). The knee injection will be given once every 12 weeks over two years for a total of eight knee injections. How well each participant tolerates each injection and all the injections over time will be assessed. The safety of getting a knee injection every 12 weeks will be assessed by collecting reported adverse effects, knee examinations, and clinical laboratory tests. Participants will complete questionnaires, X-ray, MRIs, and bone density tests as part of this study.

DETAILED DESCRIPTION:
This study was a two-year stratified and block-randomized double-blind, placebo controlled clinical trial of the effect of intra-articular triamcinolone 40 mg injectable suspension, administered every 3 months over two years (for a total of 8 doses). The randomization was stratified by the baseline radiographic severity of knee OA (Kellgren and Lawrence grade of 2 or 3) and gender. An interim analysis would have been conducted after the first half of participants has completed the trial. This interim analysis would have allowed the trial to be stopped early for either success or futility, or allow the trial to continue if neither success nor futility has been established. However, the plan for interim analysis was eliminated with the support of the DSMB because of feasibility issues for completing cartilage measurements contemporaneously and because early trial cessation would preclude analysis of informative secondary outcomes. The primary structural outcome objective in this study was cartilage volume loss; secondary structural outcomes included peri-articular bone marrow lesions (BML), tibial peri-articular bone density ratio (paBMD). The primary clinical outcome objective was the pain domain of the WOMAC© LK3.1; secondary clinical outcomes included WOMAC© LK3.1 stiffness and function scores and physical function tests.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, Age ≥ 45 years
* Chronic knee discomfort based on affirmative response to the question "During the past 12 months, have you had any pain, aching, or stiffness in or around your knee(s) on most days for at least one month?"
* Baseline (Month 0) Pain score >2 on at least one of the WOMAC weight-bearing pain questions; and total weight-bearing pain score <8
* Tibiofemoral or patellofemoral OA on posterior-anterior weight-bearing semi-flexed or lateral knee radiographs with severity equivalent to Kellgren and Lawrence grade 2 or 3
* Evidence of synovitis on ultrasound at screening
* Clinical examination confirming knee pain or discomfort referable to the knee joint
* Prepared to discontinue NSAID(s)/analgesic(s) for 2 days prior to each assessment

Exclusion Criteria:

* Prior septic (study) knee joint
* Prior reconstructive surgery in the study knee
* Prior osteonecrosis (avascular necrosis of bone)
* Chronic use of oral corticosteroids; knee intra-articular corticosteroid injection within 3 months of Month 0 (baseline) visit
* Ongoing use of doxycycline, indomethacin, glucosamine and/or chondroitin; or use of these within 2 months of Screening visit
* Evidence of other inflammatory joint disease (e.g., gout, CPPD)
* Serious medical conditions or impairments that, in the view of the investigator, would obstruct their participation in the trial such as uncontrolled diabetes, uncontrolled hypertension, opiate dependency
* Plan to permanently relocate from the region, or take an extended vacation for greater than 3 months during the trial period
* Planned arthroscopy and/or arthroplasty in the study knee.
* Any contra-indication to having an MRI
* Inability to speak or comprehend English

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E. McAlindon, MD, MPH, Principal Investigator — Tufts Medical Center / Division of Rheumatology
Locations (2):
- United States (2):
  - Tufts Medical Center / Division of Rheumatology, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McAlindon TE, LaValley MP, Harvey WF, Price LL, Driban JB, Zhang M, Ward RJ. Effect of Intra-articular Triamcinolone vs Saline on Knee Cartilage Volume and Pain in Patients With Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2017 May 16;317(19):1967-1975. doi: 10.1001/jama.2017.5283. PMID 28510679

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Chloride: Sodium chloride injection will be given into the study knee once every 12 weeks for a total of 8 injections.
  0.9% Sodium Chloride Injection as Placebo: Sodium chloride injection will be given into the study knee once every 12 weeks for a total of 8 injections.
Period: Overall Study
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone Acetonide | Sodium Chloride | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 57 | 107
  >=65 years | 20 | 13 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (8.3) | 57.2 (7.6) | 58.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 33 | 32 | 65
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Cartilage Thickness in the Index Compartment (Compartment With the Most Damage)
Description: Mean cartilage thickness was measured on knee MRI (Philips Achieva X-Series 3.0 Tesla scanner). Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Triamcinolone Acetonide 40mg: All participants received 40 mg of triamcinolone acetonide into the study knee joint every 12 weeks for a total of 8 injections.
- 0.9% Sodium Chloride: All participants received 0.9% Sodium chloride injection given into the study knee once every 12 weeks for a total of 8 injections.
Arm/Group | Triamcinolone Acetonide 40mg | 0.9% Sodium Chloride
Number analyzed (Participants) | 70 | 70
mm | -0.21 [-0.29 to -0.14] | -0.10 [-0.16 to -0.04]

2. Primary Outcome: Change in Knee Pain Severity During the Past 48 Hours From the WOMAC LK3.1 Pain Score Questionnaire.
Description: Pain subscale score was calculated from patient's responses on the Western Ontario and McMaster Universities Osteoarthritis Index Likert-type 3.1 Questionnaire. The questionnaire includes 24 items divided into 3 subscales, Pain, Stiffness, Physical Function. Only the Pain subscale score was used for this outcome measure. The Pain subscale consists of five items, each ranging from 0 to 4, making the total Pain subscore 0 to 20. Higher scores represent higher levels of pain, whereas lower scores represent lower levels of pain.
  Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
units on a scale | -1.2 [-1.9 to -0.6] | -1.9 [-2.5 to -1.2]

3. Secondary Outcome: Change in Volume of Peri-articular Bone Marrow Lesions Measured on Knee MRI.
Description: Change in volume of peri-articular bone marrow lesions measured on knee MRI on the log scale. Missing data were imputed.
Time Frame: Baseline to 2 years.
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: log mm^3
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
log mm^3 | 0.9 [-0.3 to 2.1] | 1.1 [-0.3 to 2.6]

4. Secondary Outcome: Change in Effusion Volume Measured on Knee MRI.
Description: Change in effusion volume measured on knee MRI on the log scale. Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: log mm^3
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
log mm^3 | -0.1 [-0.4 to 0.3] | -0.3 [-0.6 to -0.1]

5. Secondary Outcome: Change in Area of Denudation Measured on Knee MRI in the Index Compartment (Compartment With the Most Damage).
Description: Change in area of denudation measured on knee MRI in the index compartment (compartment with the most damage). Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: mm^2
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
mm^2 | 0.4 [0.1 to 0.8] | 0.4 [0.2 to 0.7]

6. Secondary Outcome: Change in Volumetric Cartilage Damage Index (CDI) Measured on Knee MRI in the Index Compartment (Compartment With the Most Damage).
Description: Change in volumetric cartilage damage index (CDI) measured on knee MRI in the index compartment (compartment with the most damage). Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: mm^3
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
mm^3 | -133.7 [-177.4 to -89.9] | -72.4 [-114.2 to -30.7]

7. Secondary Outcome: Change in Function Severity During the Past 48 Hours From the WOMAC LK3.1 Function Score Questionnaire.
Description: Physical Function subscale score was calculated from patient's responses on the Western Ontario and McMaster Universities Osteoarthritis Index Likert-type 3.1 Questionnaire. The questionnaire includes 24 items divided into 3 subscales, Pain, Stiffness, Physical Function. Only the Physical Function subscale score was used for this outcome measure. The Physical Function subscale consists of 17 items, each ranging from 0 to 4, making the total Function subscore 0 to 68. Higher scores represent higher levels of difficulty performing daily activities, whereas lower scores represent lower levels of difficulty performing daily activities.
  Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
units on a scale | -4.1 [-7.4 to -0.8] | -5.1 [-8.1 to -2.2]

8. Secondary Outcome: Change in Knee Stiffness During the Past 48 Hours From the WOMAC LK3.1 Stiffness Score Questionnaire.
Description: Stiffness subscale score was calculated from patient's responses on the Western Ontario and McMaster Universities Osteoarthritis Index Likert-type 3.1 Questionnaire. The questionnaire includes 24 items divided into 3 subscales, Pain, Stiffness, Physical Function. Only the Stiffness subscale score was used for this outcome measure. The Stiffness subscale consists of two items, each ranging from 0 to 4, making the total Stiffness subscore 0 to 8. Higher scores represent higher levels of stiffness, whereas lower scores represent lower levels of stiffness.
  Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
units on a scale | -0.6 [-1.1 to -0.1] | -0.5 [-1.0 to 0]

9. Secondary Outcome: Change in Patient's Global Assessment (Visual Analogue Scale).
Description: The response to the question, "Considering all the ways your knee affects you, how much pain are you having today?", was measured and the change in the scoring was evaluated. The Patient's Global Assessment (PGA) is measured on a scale of 0 to 100 millimeters. Higher scores represent a higher level of disease activity or a worse global health. Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
mm | -2.7 [-11.9 to 6.6] | -7.6 [-15.4 to 0.2]

10. Secondary Outcome: Change in Time to Complete a Twenty-meter Walk.
Description: Change in time (seconds) to complete a twenty-meter walk. Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
seconds | -0.3 [-1.0 to 0.4] | 0.1 [-0.6 to 0.9]

11. Secondary Outcome: Change in Time to Complete 5 Chair Stands.
Description: Change in time (seconds) to complete 5 chair stands. Missing data were imputed.
Time Frame: Baseline to 2 years
Population: All individuals were included in analysis, which was performed on multiply imputed data.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Number analyzed (Participants) | 70 | 70
seconds | -1.1 [-3.5 to 1.2] | -1.2 [-3.6 to 1.1]

ADVERSE EVENTS:
Arm/Group | Triamcinolone Acetonide | Sodium Chloride
Serious Adverse Events (participants affected / at risk) | 15/70 | 27/70
Other Adverse Events (participants affected / at risk) | 48/70 | 60/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triamcinolone Acetonide (N=70) | Sodium Chloride (N=70)
Asthma excerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Liver and bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Hemorrhoid (Gastrointestinal disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Foot surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Blood clot in leg (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fractured humerus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Benign cyst surgical removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Melanoma surgical removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
fever (General disorders) | 0 (0) | 1 (1)
Infra-hisian block (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Achilles Tendon tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suddden Death (General disorders) | 0 (0) | 1 (1)
Cholesteatoma (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Appendiceal mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Metformin toxicity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alcohol withdrawal (Nervous system disorders) | 0 (0) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Metastatic Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ductal carcinoma insitu (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Weakness and chest pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triamcinolone Acetonide (N=70) | Sodium Chloride (N=70)
Dog bites on left wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dysphagia and Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Increase in atorvastatin dosage (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastrophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 6 (6) | 10 (10)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3)
Chronic Kidney Disease-Stage III (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 1 (1)
Broken Toe (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0)
Bladder infections (Infections and infestations) | 0 (0) | 1 (1)
Swollen left knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus Infection (Infections and infestations) | 3 (4) | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chest cold (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 12 (13)
Right foot pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Left (index) knee sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
thyroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Walking pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Anxiety attack (Psychiatric disorders) | 1 (1) | 0 (0)
Fractured rib (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Bruised ribs (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shingles (Infections and infestations) | 2 (2) | 0 (0)
Reaction to shingle vaccine (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Established hypertension (Vascular disorders) | 0 (0) | 2 (2)
Transient hypertension (Vascular disorders) | 1 (1) | 0 (0)
Sprained wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
Increased neck and facial muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Perimenopause and ovarian cyst flare (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bursitis in hips (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Ankle sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Left foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stomach virus (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Stomach pain and vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Closed head injury with scalp laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infective conjunctivitis (Infections and infestations) | 0 (0) | 1 (2)
Head cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Diffuse joint pain (Nervous system disorders) | 0 (0) | 1 (1)
Herniated Disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chipped Tooth (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 2 (2)
Gout flare in big toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Erythema-facial (Immune system disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Left ankle pain and swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (2) | 2 (2)
Syncope (Cardiac disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Yeast Infection (Infections and infestations) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Cold symptoms (General disorders) | 8 (8) | 4 (5)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain - abdominal and lower back (General disorders) | 0 (0) | 1 (1)
Rhinovirus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Left (index) knee tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Infections and infestations) | 1 (1) | 2 (3)
Injection site pain (General disorders) | 4 (4) | 2 (2)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Benign Prostatic hyperplasia (Renal and urinary disorders) | 0 (0) | 1 (1)
Left ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Right (index) knee joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Body pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Insomnia and anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Right knee burning sensation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Superficial knee scrape & laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 3 (3) | 1 (1)
Right (non-index) hamstring strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parasite (nematode) in left eye (Infections and infestations) | 0 (0) | 1 (1)
Left arm contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Torn ACL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Right (index) knee joint discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Locked right (index) knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sciatica (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Sciatica flare (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pre-cancerous mole-left forearm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Post-surgical incision site infection - left forearm (General disorders) | 0 (0) | 1 (1)
Polycythemia vera (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Torn meniscus - left knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Allergic bronchitis (Immune system disorders) | 1 (1) | 0 (0)
Hiatal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Left heel fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cellulitis - right hand (Infections and infestations) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Right (index) knee pain & swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left (index) knee swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Strained muscle - back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Uterine fibroid (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome - bilateral hands (Nervous system disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Knee contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dislocated right middle finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Left shoulder strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Synovial cyst - lumbar spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pain - right shoulder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rotator cuff tear - right shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Right leg pain (General disorders) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Bruising - left wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Plan for interim analysis was eliminated with the support of the DSMB because of feasibility issues for completing cartilage measurements contemporaneously and because early trial cessation would preclude analysis of informative secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No